CLINICAL TRIAL: NCT00777218
Title: Cognitive Side Effects of Commonly Prescribed Medications in Pediatric Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment criteria was too challenging and Investigators changed Institutions
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-185
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Propranolol; Zonisamide; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: propranolol
- 2 (Active Comparator)
  Interventions: Drug: zonisamide
- 3 (Active Comparator)
  Interventions: Drug: topiramate

INTERVENTIONS:
Drug: propranolol — standard pediatric doses, based on body weight
  Other Names: Inderal
  Arms: 1
Drug: zonisamide — standard pediatric dosages, based on body weight
  Other Names: Zonegran
  Arms: 2
Drug: topiramate — standard pediatric dosages, based on body weight
  Other Names: Topamax
  Arms: 3

SUMMARY:
The purpose of this study is to determine if there are significant differences in the side effects related to memory, repetition and recall among these three drugs when used in a pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of migraine with and without aura or chronic daily headache as defined by IHS
* subjects must between the age of 8-17 (inclusive)

Exclusion Criteria:

* diagnosis of tension-type headache or cluster headache

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Record if memory, repetition or recall was impaired by subject during specific time frame on medication. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: J. I. Lopez, MD, Principal Investigator — University of South Alabama Department of Neurology
Locations (1):
- University of South Alabama Department of Neurology, Mobile, Alabama, United States